CLINICAL TRIAL: NCT01799512
Title: Randomized Evaluation of Glycaemic Control in the Medical Intensive Care Unit Using Continuous Glucose Monitoring (REGIMEN Trial)
Brief Title: Glucose Control in the ICU Using Continuous Glucose Monitoring
Acronym: REGIMEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Christophe De Block, MD PhD, University Hospital, Antwerp
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REGIMEN
Record Dates: First submitted 2013-02-20; First posted 2013-02-26 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Critical Illness
Keywords: medical ICU patients; APACHE-II score ≥20
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- real-time continuous glucose monitoring (Experimental): real-time continuous glucose monitoring: Use will be made of the online real-time (RT) monitoring facility of the GlucoDay® (a continuous glucose monitoring (CGM)system). This will allow immediate adaptation of the insulin dose in order to maintain values within an optimal range.
  The same IV insulin infusion protocol will be used in the experimental and the active comparator group (adapted Yale protocol).
  When glycaemic changes of >25 mg/dl per 30 minutes are observed from the RT-CGM - GlucoDay data, this will be checked by measuring arterial blood glucose and the insulin infusion rate will be adapted according to the adapted Yale protocol.
  Interventions: Device: experimental: real-time continuous glucose monitoring
- blinded continuous glucose monitoring (Active Comparator): In the active comparator group the same continuous glucose monitoring device (GlucoDay) will be used in a blinded fashion. Glucose data will be analysed retrospectively.
  IV insulin infusion will be adapted according to arterial blood glucose values, using the adapted Yale protocol.
  Interventions: Device: Active comparator: blinded continuous glucose monitoring

INTERVENTIONS:
Device: experimental: real-time continuous glucose monitoring
  Other Names: RT-CGM using the GlucoDay device (A. Menarini, Italy)
  Arms: real-time continuous glucose monitoring
Device: Active comparator: blinded continuous glucose monitoring
  Arms: blinded continuous glucose monitoring

SUMMARY:
Stress hyperglycemia occurs in 50-85% of patients admitted to a medical intensive care unit (MICU) and is associated with increased morbidity and mortality. However, randomized controlled trials examining the effects of strict glycemic control demonstrated conflicting results. A common finding in these trials was the high risk of hypoglycaemia.

This randomized controlled trial evaluates the impact of real-time continuous glucose monitoring (RT-CGM) on glycemic control and risk of hypoglycemia in severely ill MICU patients with an APACHE-II (Acute Physiology and Chronic Health Evaluation II) score ≥20.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to a medical intensive care unit
* age: ≥ 18 y , < 75 y
* APACHE II (Acute Physiology and Chronic Health Evaluation II) score ≥ 20
* expected length of stay in ICU > 3 days

Exclusion Criteria:

* pregnancy
* patient with a DNR (do not reanimate) code
* surgical patient
* no informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-07; Primary Completion 2010-09 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
percentage of time that patients are in target range of glycaemia (80-110 mg/dl) | participants will be followed for 96 hours (4 days), during the first week after admission to the medical ICU
  after admission to the ICU, patients will be screened to check inclusion criteria, and CGM monitoring will commence within the first 48hrs after admission. CGM monitoring will be performed during 96 hours (4 days), during the first week after admission to the medical ICU

SECONDARY OUTCOMES:
percentage of time that patients are in hypoglycaemic range | participants will be followed for 96 hours (4 days), during the first week after admission to the medical ICU
  after admission to the ICU, patients will be screened to check inclusion criteria, and CGM monitoring will commence within the first 48hrs after admission. CGM monitoring will be performed during 96 hours (4 days), during the first week after admission to the medical ICU

OTHER OUTCOMES:
accuracy of continuous glucose monitoring | participants will be followed for 96 hours (4 days), during the first week after admission to the medical ICU
  error grid analysis, analysing all data of the 4 days of continuous glucose monitoring period
glycaemic fluctuations | participants will be followed for 96 hours (4 days), during the first week after admission to the medical ICU
  standard deviation of mean glucose value over 4 days, analysing all data of the 4 days of continuous glucose monitoring period
accuracy of continuous glucose monitoring | participants will be followed for 96 hours (4 days), during the first week after admission to the medical ICU
  Bland-Altman bias plot will be evaluated, analysing all data of the 4 days of continuous glucose monitoring period
accuracy of continuous glucose monitoring | participants will be followed for 96 hours (4 days), during the first week after admission to the medical ICU
  mean absolute error and mean relative error will be evaluated, analysing all data of the 4 days of continuous glucose monitoring period
glycaemic fluctuations | participants will be followed for 96 hours (4 days), during the first week after admission to the medical ICU
  MAGE (mean amplitude of glucose excursions), analysing all data of the 4 days of continuous glucose monitoring period
glycaemic fluctuations | participants will be followed for 96 hours (4 days), during the first week after admission to the medical ICU
  CONGA (continuous overlapping net glycemic action), analysing all data of the 4 days of continuous glucose monitoring period
glycaemic fluctuations | participants will be followed for 96 hours (4 days), during the first week after admission to the medical ICU
  area under curve (within target glycemia range, above target, below target) analysing all data of the 4 days of continuous glucose monitoring period
glycaemic fluctuations | participants will be followed for 96 hours (4 days), during the first week after admission to the medical ICU
  MODD: mean of daily differences; analysing all data of the 4 days of continuous glucose monitoring period

CONTACTS AND LOCATIONS:
Overall Officials: Christophe De Block, MD PhD, Principal Investigator — Antwerp University Hospital, Dept of Endocrinology, Diabetology & Metabolism
Locations (2):
- Belgium (2):
  - Middelheim General Hospital, Antwerp
  - Antwerp University Hospital, Edegem

REFERENCES:
- [Background] De Block C, Manuel-Y-Keenoy B, Van Gaal L, Rogiers P. Intensive insulin therapy in the intensive care unit: assessment by continuous glucose monitoring. Diabetes Care. 2006 Aug;29(8):1750-6. doi: 10.2337/dc05-2353. PMID 16873775
- [Background] De Block C, Manuel-y-Keenoy B, Rogiers P, Jorens P, Van Gaal L. Glucose control and use of continuous glucose monitoring in the intensive care unit: a critical review. Curr Diabetes Rev. 2008 Aug;4(3):234-44. doi: 10.2174/157339908785294460. PMID 18690906
- [Background] Goldberg PA, Siegel MD, Sherwin RS, Halickman JI, Lee M, Bailey VA, Lee SL, Dziura JD, Inzucchi SE. Implementation of a safe and effective insulin infusion protocol in a medical intensive care unit. Diabetes Care. 2004 Feb;27(2):461-7. doi: 10.2337/diacare.27.2.461. PMID 14747229
- [Background] Shetty S, Inzucchi SE, Goldberg PA, Cooper D, Siegel MD, Honiden S. Adapting to the new consensus guidelines for managing hyperglycemia during critical illness: the updated Yale insulin infusion protocol. Endocr Pract. 2012 May-Jun;18(3):363-70. doi: 10.4158/EP11260.OR. PMID 22138078
- [Background] Holzinger U, Warszawska J, Kitzberger R, Wewalka M, Miehsler W, Herkner H, Madl C. Real-time continuous glucose monitoring in critically ill patients: a prospective randomized trial. Diabetes Care. 2010 Mar;33(3):467-72. doi: 10.2337/dc09-1352. Epub 2009 Dec 10. PMID 20007948
- [Derived] De Block CE, Gios J, Verheyen N, Manuel-y-Keenoy B, Rogiers P, Jorens PG, Scuffi C, Van Gaal LF. Randomized Evaluation of Glycemic Control in the Medical Intensive Care Unit Using Real-Time Continuous Glucose Monitoring (REGIMEN Trial). Diabetes Technol Ther. 2015 Dec;17(12):889-98. doi: 10.1089/dia.2015.0151. Epub 2015 Aug 25. PMID 26305390